CLINICAL TRIAL: NCT06816212
Title: Correlation Between CEUS Identification of Hepatic Nodular Perfusion Disorders on CE-MRI and Hepatic Malignant Lesions: a Prospective Multicenter Study
Brief Title: Correlation Between CEUS Identification of Nodular HPD on CE-MRI and Hepatic Malignant Lesions
Status: Enrolling by invitation | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-0104
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Hepatic Malignant Tumors; Hepatic Perfusion Disorders
Keywords: Hepatic malignant tumors; US-MRI image fusion; Contrast-Enhanced Ultrasound; quantitative analyses; Hepatic perfusion disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Benign nodular hepatic perfusion disorders: Perform contrast-enhanced ultrasound examination on the benign nodular hepatic perfusion disorders and analyze the images
- Hepatic malignant lesions: Perform contrast-enhanced ultrasound examination on the hepatic malignant lesions and analyze the images

SUMMARY:
Hepatic malignant tumors are a category of diseases with high incidence and mortality rates worldwide, including various types such as primary hepatocellular carcinoma (HCC), intrahepatic cholangiocarcinoma (ICC), and liver metastases. With the advancement of imaging technology, the number of hepatic perfusion disorders (HPD) detected in high-risk population screening and follow-up has gradually increased. However, the imaging manifestations of these HPD are highly heterogeneous, and the imaging features of some benign lesions (such as post-treatment inflammatory reactions, arterioportal shunts, hyperplastic nodules, focal fat deposition or fibrotic nodules) overlap with those of malignant lesions, posing a challenge to accurate diagnosis. Therefore, how to improve the ability to distinguish the benign and malignant nature of HPD based on multimodal imaging technology and optimize the follow-up management of high-risk populations has significant clinical value.

DETAILED DESCRIPTION:
Hepatic malignant tumors, including hepatocellular carcinoma (HCC), intrahepatic cholangiocarcinoma (ICC), and liver metastases, represent a significant global health burden due to their high incidence and mortality rates. With advancements in imaging techniques, the detection of hepatic perfusion disorders (HPD) in high-risk populations during screening and follow-up has increased. However, the imaging characteristics of HPD lack distinct heterogeneity, and certain benign lesions-such as post-treatment inflammatory reactions, arterioportal shunts, hyperplastic nodules, focal fat deposition, or fibrotic nodules-may exhibit overlapping imaging features with malignant lesions, posing a challenge for accurate diagnosis.

Contrast-enhanced magnetic resonance imaging (CE-MRI) is a key modality for evaluating hepatic nodules. However, it has limitations in differentiating non-typical enhancement patterns of lesions, such as metastases with minimal microvascular invasion, as well as non-specific nodules in cirrhotic backgrounds. Contrast-Enhanced Ultrasound (CEUS), with its unique ability to provide real-time dynamic assessment of tumor perfusion, is increasingly recognized as a valuable tool for hepatic lesion evaluation. Compared to CE-MRI, CEUS offers superior temporal resolution and lower costs, particularly in early post-treatment efficacy assessment, hemodynamic evaluation, and differentiation of residual viable tumor tissue from post-treatment changes. Moreover, ultrasound-MRI fusion imaging enhances the detection of small hepatic lesions, while CEUS quantitative analysis allows for the evaluation of tumor microvascular parameters to predict early malignant transformation. These advancements provide a more reliable approach for identifying malignant HPD using CEUS-based techniques.

This multicenter, prospective study aims to integrate ultrasound-MRI fusion imaging and CEUS quantitative analysis to improve the precise identification of early malignant lesions within nodular HPD detected on CE-MRI. Additionally, this study seeks to establish high-level evidence supporting the use of CEUS with ultrasound-MRI fusion for accurate localization and characterization of malignant lesions. Ultimately, the findings will contribute to the optimization of surveillance strategies for high-risk populations, including individuals at risk for hepatocellular carcinoma and other malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

* Prospective cohort patients voluntarily sign the informed consent form.
* Patients with a history of malignant tumors, CE-MRI indicated the presence of HPD in the liver.
* The shape of HPD is nodular.
* The diameter of HPD is greater than 10mm.
* The main large vessels in the liver are clearly displayed in the MRI.

Exclusion Criteria:

* Patients who unable to complete imaging examinations, such as severe cardiac insufficiency, severe renal insufficiency, hypersensitivity to contrast agents or adverse reactions to them, etc.
* Patients with the history of extensive liver resection or liver transplantation.
* Patients whose abdomen with abundant intestinal gas.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with nodular hepatic perfusion disorders
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2025-02-10 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy | 2 years
  The diagnostic model correctly distinguish between hepatic malignant lesions and benign nodular hepatic perfusion disorders.
Correlation | 2 years
  Correlation between nodular HPD and hepatic malignant lesions
False negative rate | 2 years
  The probability of misdiagnosing malignant liver lesions as benign nodular HPD by CE-MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ultrasound, Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
The data cannot be shared because of ethical restrictions regarding human participant data.